CLINICAL TRIAL: NCT05495932
Title: Mepolizumab Pharmacokinetics Among Patients With Severe Asthma: Protocol for a Case Control Study Comparing Clinical Responders Versus Non Responders
Brief Title: Mepolizumab Pharmacokinetics Among Patients With Severe Asthma
Acronym: CESAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0035; 2022-A00982-41 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-01

CONDITIONS: Asthma
Keywords: Severe asthma; Mepolizumab; Biologics; Response; Pharmacokinetics
MeSH Terms: conditions — Asthma | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Case-control study including adult patients with severe asthma successfully treated with mepolizumab for at least 24 weeks, and then divided into two groups at inclusion : responders and non-responders according to the results of blood samples taken at inclusion, 1 month and 6 months during study follow-up
  The clinical criteria used to define a complete response to mepolizumab are : Reduction of maintenance corticotherapy > 50% reduction OR dose >5mg/day; Reduction of exacerbation rate by > 50%; ACQ-6 score < 1.5 and no increase in score > 0.5 since enrolment Patients lacking any one of the previous criteria are classified as non-responders.
  Clinical response criteria are evaluated at each study visit, and the final classification at 6 months post-inclusion determines study groups to be matched and compared during statistical analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eligible patients (Experimental)
  Interventions: Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: blood sample — blood sample taken to measure serum mepolizumab concentration at baseline, 1 month and 6 months during study follow-up

SUMMARY:
Asthma is a chronic disease characterized by inflammation and obstruction of the airways. Identification of the mechanisms of action of corticosteroids has made it possible to define the type 2 inflammation present in nearly 80% of patients with asthma.

Monoclonal antibodies (MAb) in severe asthma target type-2 inflammation. Mepolizumab is a humanized IgG1 (immunoglobulin gamma-1) kappa subclass monoclonal antibody directed specifically against interleukin 5 (IL-5). It acts specifically on eosinophil homeostasis, with IL-5 being a key interleukin in eosinophil maturation.

The investigators propose to measure the concentrations of mepolizumab in the serum of asthmatic patients treated with this mAb. The investigators hypothesize that the individual pharmacokinetics (PK) of mepolizumab may differ between clinical responders and non-responders.

DETAILED DESCRIPTION:
Asthma is a chronic disease characterized by inflammation and obstruction of the airways. Understanding the biological effects of the corticosteroids allowed to identify and to define the type 2 inflammation present in nearly 80% of patients with asthma.

Monoclonal antibodies (MAb) in severe asthma target type-2 inflammation. Mepolizumab is a humanized IgG1 kappa subclass monoclonal antibody directed specifically against interleukin 5 (IL-5). It acts specifically on eosinophil homeostasis, since IL-5 is a key interleukin in eosinophil maturation.

Poor MAb responses can hypothetically arise in situations of poor treatment compliance. And after excluding the latter, several biological mechanisms have been mentioned: i) insufficient bioavailability of the MAb to reach the eosinophils of the bronchial compartment; ii) he development of autoimmunity with the formation of circulating immune complexes; and iii) immunization against mepolizumab, with the formation of neutralizing anti-drug antibodies (ADA).

ADA were detected in up to 20% of a treated population and were rarely neutralizing.

Interestingly, these ADA could also be detected in naïve populations, suggesting a possible cross-immunization related to previous exposure to MAbs and/or to insufficient assay specificity. In any case, all three possibilities have a common outcome, i.e. decreased circulating concentrations of the MAb in the blood.

The investigators propose to measure the concentrations of mepolizumab in the serum of asthmatic patients treated with this mAb. The investigators hypothesize that the individual pharmacokinetics (PK) of mepolizumab may differ between clinical responders and non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age: 18 years old
* History of severe asthma diagnosed by a physician (according to Global Initiative for Asthma (GINA) criteria)
* Subject on a combination of high-dose (ICS equivalent to 1000 μg beclomethasone) and medium dose inhaled corticosteroid and long acting beta-agonists at least 12 months before inclusion
* Treatment with mepolizumab in line with the Marketing Authorization
* Having received at least 6 doses of mepolizumab (monthly subcutaneous administration)
* Documented initial clinical response to mepolizumab

Exclusion Criteria:

* Other respiratory diseases
* Potential interference from another study
* Immunosuppressive treatment (i.e methotrexate, polyvalent immunoglobulins, other monoclonal antibody for other condition such as cancer; oral and/or inhaled corticosteroids are allowed)
* Populations protected according to the French public health code
* Patient is unavailable, unable or unwilling to attend future visits
* Non-beneficiary of the French national health insurance system
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Mepolizumab serum concentration | 1 month
  The primary outcome is the change in trough concentration of mepolizumab in serum at 1-month post-enrolment. Mepolizumab serum concentration will be determine by ELISA

SECONDARY OUTCOMES:
Mepolizumab serum concentration | 6 months
  Mepolizumab serum concentration will be determine by ELISA.
Complete blood cell count at 1 month | 1 month
  comparison of number and % of eosinophils, basophils, neutrophils between responders and non-responders at baseline and 1-month
Complete blood cell count at 6 months | 6 months
  comparison of number and % of eosinophils, basophils, neutrophils between responders and non-responders for the six-month follow-up period
Comparison of lung function by airway obstruction | 6 months
  To describe the degree of airway obstruction, forced expiratory volume in one second (FEV1) and forced vital capacity will be measured using spirometry. The quantitative variables FEV1 and FEV1/FVC (Forced Vital Capacity) will be compared between responders and non-responders for the six-month follow-up period
Comparison of asthma control by ACQ-6 score | 6 months
  Asthma control in terms of symptoms will be assessed by the six-item Asthma Control Questionnaire (ACQ-6). The ACQ-6 scores will be compared between responders and non-responders for the six-month follow-up period.
  Patients are asked to recall how their asthma has been during the previous week by responding to one bronchodilator use question and 5 symptom questions.
  Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-6 score is the mean of the responses.
  A score of 1.5 or more on the 6-item Asthma Control Questionnaire (ACQ-6) indicates that a patient has inadequate asthma control.
Comparison of chronic rhinosinusitis by SNOT-22 score | 6 months
  The sino-nasal outcomes for chronic rhinosinusitis will be assessed by the 22-item sino-nasal outcome test (SNOT-22). The SNOT-22 scores will be compared between responders and non-responders for the six-month follow-up period.
  The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110. Higher scores indicate poorer outcomes.
Comparison of exacerbation rate | 6 months
  Number, dates, and severity of exacerbations as defined by the Global Asthma Initiative (GINA) will be collected throughout the follow-up period. The number of exacerbations, the exacerbations rate and the number of days not exacerbating will be compared between responders and non-responders.
Number of days alive and not exacerbating | 6 months
Comparison of change in oral corticosteroid | 6 months
  Oral corticosteroid use will be collected throughout the follow-up period. The % decrease of the initial corticosteroid therapy will be compared between responders and non-responders at 6 months.
Presence/absence of a >50% reduction in exacerbation rate | 6 months
Presence/absence of monoclonal antibody switching | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie GAMEZ, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (2):
- France (2):
  - university Hospital of Montpellier, Montpellier, France
  - University Hospital of Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Yes
The general goal is to make the study data available to interested researchers as well as to provide proof of transparency for the study.
  Data will be made available to persons who address a reasonable request to the study director.
  Individual participant data (and an accompanying data dictionary) will be de-identified and potentially further cleaned or aggregated as the investigators deem necessary to protect participant anonymity.
  The following will also be made available to the public at https://osf.io/a5cdg/ as soon as feasible:
  * The study protocol (will preferably be published in a journal; alternatively, it can be posted to https://osf.io/a5cdg/);
  * Participant information materials;
  * The paper form for the eCRF;
  * The data sharing plan.
Supporting Information: Study Protocol
Time Frame: Datasets that underlie the results reported in the article (text, tables, figures, and appendices) can be requested after the publication process has been completed.
Access Criteria: The conditions under which members of the public will be granted access to datasets are:
  * The data will be used/examined in a not-for-profit manner;
  * The data will not be used in an attempt to identify a participant or group of participants;
  * The user does not work for a private insurance company;
  * The data will not be used in support of any kind of private insurance policy or health penalties;
  * The data will be used/examined for the advancement of science/teaching while respecting participant/patient privacy and rights;
  * The user will state why they wish to access the data.
  * If the data do not fulfil the requirements of the reference methodology (MR-001) (ex: data about religion, etc.), the appropriate CNIL (National Commission for Computing and Liberties) approval has to be obtained by the user.
  * If the data will be used outside the European Union, standard contractual clauses have to be signed between Montpellier University Hospital and the user before sharing data.
URL: https://osf.io/a5cdg/